CLINICAL TRIAL: NCT02103764
Title: The Effectiveness of Cyclic Desogestrel Therapy for Abnormal Uterine Bleeding Associated With Anovulation: a Non-inferiority Double Blinded Randomized Control Trial
Brief Title: Efficacy of Cyclic DSG Compared With Cyclic MPA for the Treatment of Anovulatory DUB
Acronym: SI-AUB-RCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Manee Rattanachaiyanont, Department of Obstetrics and Gynecology, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSG-SIAUB
Record Dates: First submitted 2014-02-18; First posted 2014-04-04 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Dysfunctional Uterine Bleeding
Keywords: Anovulatory Dysfunctional Uterine Bleeding; cyclic desogestrel; cyclic medroxyprogesterone acetate; lipid metabolism; glucose metabolism; endometrial histology changing
MeSH Terms: conditions — Metrorrhagia | interventions — Desogestrel; Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desogestrel (Experimental): Desogestrel Dosage form : Desogestrel 150 mcg/capsule Dosage : 150 mcg/day Frequency : 1 capsule/day before bed time Duration: 10 day/month
  Interventions: Drug: Desogestrel
- Medroxyprogesterone acetate (Active Comparator): Medroxyprogesterone acetate Dosage form : 10 mg./capsule Dosage : 10 mg./day Frequency : 1 capsule/day before bed time Duration : 10 day/month
  Interventions: Drug: Medroxyprogesterone acetate

INTERVENTIONS:
Drug: Desogestrel — Desogestrel Dosage form : Desogestrel 150 mcg/capsule Dosage : 150 mcg/day Frequency : 1 capsule/day before bed time Duration: 10 day/month
  Other Names: Cerazette
  Arms: Desogestrel
Drug: Medroxyprogesterone acetate — Medroxyprogesterone acetate Dosage form : 10 mg./capsule Dosage : 10 mg./day Frequency : 1 capsule/day before bed time Duration : 10 day/month
  Other Names: Provera
  Arms: Medroxyprogesterone acetate

SUMMARY:
The objectives of the present study is to determine the effectiveness of cyclic desogestrel (DSG) compared with cyclic medroxyprogesterone acetate for the treatment of anovulatory dysfunctional uterine bleeding (DUB) in the following aspects:

1. Endometrial histopathology changes
2. Menstrual cycle control.

DETAILED DESCRIPTION:
Anovulatory dysfunctional uterine bleeding (DUB) is the most common cause of abnormal uterine bleeding especially in postmenarcheal adolescent, perimenopausal women, patient with polycystic ovary syndrome (PCOS) and in obese women. Aims of treatment in women with anovulatory DUB are to restore the natural control mechanism of endometrium (introduce normal synchronous growth, development, shedding of a structural stable endometrium) and to prevent endometrial hyperplasia. The two main treatment options are estrogen-progestin therapy and progestin therapy. Women who are sexually active and not immediately prepared to pursue pregnancy are best manage by estrogen-progestin treatment especially combined oral contraceptive pills (COCs) but in perimenopausal women, obese women or women who can't tolerate COCs or have contraindications in using COCs, cyclic progestin will be the treatment of choice. Common used progestin in anovulatory DUB is medroxyprogesterone acetate (MPA) 5-10 mg/day for 10-14 days each month. This progestin has strong progestogenic effect but has some undesirable effect such as glucocorticoid effect, mineralocorticoid effect and androgenic effect. Long term using this progestin especially in obese women or perimenopausal women who have risk for diabetes mellitus and dyslipidemia may be negative effect to glucose and lipid metabolism. DSG is the third generation progestin with no glucocorticoid, mineralocorticoid effect and low androgenic effect may be the better choice of treatment but the data of DSG in treatment of anovulatory DUB us scanty. So this study will evaluate the effect of cyclic DSG in endometrial histology changing and lipid, glucose metabolism in patient with anovulatory DUB.

Comparison : Women with anovulatory DUB are randomized into two groups, receiving a course of either cyclic DSG or cyclic MPA. The main outcome measured is to compare the effect of both interventions on endometrial histology changing.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with anovular DUB (proved by endometrial histology)
* Age > 18 yr.

Exclusion Criteria:

* Any uterine pathology that might cause abnormal uterine bleeding
* Contraindication to progestin treatment (such as breast cancer)
* Severe drug allergy towards a progestogen
* Intake of any hormonal treatment in the previous 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The change in endometrial histology | Baseline, Day 8 or 9 or 10 of treatment period in first month
  The participants are evaluated for changing of endometrial histology at day 8 or 9 or 10 of treatment period.

SECONDARY OUTCOMES:
The occurrence of withdrawal bleeding | 6 months
  To compare the occurrence of withdrawal bleeding between cyclic DSG and cyclic MPA groups.
Effect of cyclic DSG on lipid metabolism compared with cyclic MPA | 6 months
  To compare the change of total cholesterol (TC), triglyceride, HDL-C, and LDL-C between cyclic DSG and cyclic MPA groups.
Effect of cyclic DSG on glucose metabolism compared with cyclic MPA | 6 months
  To compare the change of fasting blood glucose, and fasting insulin between cyclic DSG and cyclic MPA groups.
Adverse events | At day 8 or 9 or 10 of the first cycle and 3, 6 month
  To compare the adverse events, including side effects between cyclic DSG and cyclic MPA groups.

CONTACTS AND LOCATIONS:
Overall Officials: Manee Rattanachaiyanont, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Soontrapa N, Rattanachaiyanont M, Warnnissorn M, Wongwananuruk T, Indhavivadhana S, Tanmahasamut P, Techatraisak K, Angsuwathana S. The effectiveness of desogestrel for endometrial protection in women with abnormal uterine bleeding-ovulatory dysfunction: a non-inferiority randomized controlled trial. Sci Rep. 2022 Jan 31;12(1):1662. doi: 10.1038/s41598-022-05578-0. PMID 35102226